CLINICAL TRIAL: NCT07306702
Title: Effect of Dexmedetomidine Combined With Oseltamivir Fumarate for Patient-controlled Intravenous Analgesia Following Lobectomy in Patients With Nicotine Dependence
Brief Title: Dexmedetomidine-Enhanced PCIA After Lobectomy in Nicotine-Dependent Patients
Acronym: DEX-PCIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Yu Shang, Principal Investigator, Shenyang Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYCHS6-LOB-PCIA-RCT-2023; JUH-CCP-RC-RETRO-01 (Other: Shenyang Sixth People's Hospital)
Record Dates: First submitted 2025-11-21; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain Management
MeSH Terms: interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oliceridine PCIA Alone (Active Comparator): Postoperative patient-controlled intravenous analgesia (PCIA) using oliceridine only. Reservoir 100 mL; basal 2 mL/h; bolus 0.5 mL; lockout 15 min; ~3 mL loading dose given near the end of surgery. Used for up to 48 h after lobectomy. Tramadol 50-100 mg IV permitted as rescue per protocol. No dexmedetomidine infusion.
  Interventions: Drug: Oliceridine
- Oliceridine + Low-Dose Dexmedetomidine (Experimental): Same oliceridine PCIA parameters as Arm 1, plus a continuous IV infusion of dexmedetomidine at 0.05 μg/kg/h (0.05 mcg/kg/h) for up to 48 h postoperatively. Tramadol 50-100 mg IV permitted as rescue per protocol.
  Interventions: Drug: Oliceridine; Drug: Dexmedetomidine
- Oliceridine + Standard-Dose Dexmedetomidine (Experimental): Same oliceridine PCIA parameters as Arm 1, plus a continuous IV infusion of dexmedetomidine at 0.10 μg/kg/h (0.1 mcg/kg/h) for up to 48 h postoperatively. Tramadol 50-100 mg IV permitted as rescue per protocol.
  Interventions: Drug: Oliceridine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Oliceridine — Patient-controlled intravenous analgesia (PCIA) after VATS lobectomy using oliceridine only. 100-mL reservoir; basal rate 2 mL/h; 0.5-mL bolus; 15-min lockout; ~3-mL loading near end of surgery; used for up to 48 h. Tramadol 50-100 mg IV permitted as rescue per protocol.
Drug: Dexmedetomidine — Continuous IV infusion as an adjuvant to the oliceridine PCIA per group assignment for up to 48 h: 0.05 μg/kg/h in Arm 2 or 0.10 μg/kg/h in Arm 3. Infusion may be held for HR <50 bpm or MAP <65 mmHg per protocol.
  Arms: Oliceridine + Low-Dose Dexmedetomidine; Oliceridine + Standard-Dose Dexmedetomidine

SUMMARY:
This randomized, double-blind, controlled clinical trial evaluates whether adding dexmedetomidine to an oliceridine-based patient-controlled intravenous analgesia (PCIA) regimen can improve postoperative pain control and tolerability after video-assisted thoracoscopic lobectomy in adults with high nicotine dependence (Fagerström score ≥6). A total of 102 participants are allocated 1:1:1 into three groups: (1) oliceridine PCIA alone; (2) oliceridine PCIA plus low-dose dexmedetomidine (0.05 μg/kg/h); or (3) oliceridine PCIA plus standard-dose dexmedetomidine (0.1 μg/kg/h). PCIA solutions are prepared to 100 mL, delivered with a basal rate of 2 mL/h, a 0.5-mL bolus, and a 15-minute lockout; a small loading dose is given near the end of surgery. Tramadol is permitted as rescue analgesia per protocol.

The primary objectives are to compare postoperative pain intensity at rest and with movement and overall patient satisfaction within 48-72 hours after surgery. Secondary objectives include sedation level, negative affect (anxiety/depression) scores, comfort and functional recovery scales, effective PCIA presses, rescue analgesic use, and safety outcomes (nausea/vomiting, shivering, bradycardia, hypotension, hypoxemia, and respiratory depression). Outcomes are assessed at approximately 4, 8, 12, 24, and 48 hours after surgery, with a satisfaction survey at 72 hours.

The investigators hypothesize that oliceridine PCIA combined with dexmedetomidine-particularly at 0.1 μg/kg/h-will reduce movement-related pain, decrease rescue opioid needs and PCIA presses, improve mood and comfort scores, and maintain acceptable hemodynamic and respiratory safety compared with oliceridine alone.

DETAILED DESCRIPTION:
Adults scheduled for first-time thoracoscopic lobectomy at two centers are screened preoperatively; key exclusions include significant conduction abnormalities, severe organ dysfunction, inability to use PCIA, or recent exposure to α2-agonists/opioids that could confound results. After surgery, participants are randomized to one of three masked PCIA regimens. Study personnel, patients, and outcome assessors remain blinded. Standardized anesthetic and postoperative care pathways are followed. Pain (rest/movement visual analog scales), sedation (Ramsay), mood (self-rating anxiety/depression), comfort/function scales, and adverse events are recorded at prespecified time points through 48 hours; patient satisfaction is collected at 72 hours. Data are analyzed with appropriate parametric/non-parametric tests for continuous variables and χ²/Fisher's exact tests for categorical outcomes, with two-sided α=0.05.

ELIGIBILITY:
Inclusion Criteria

* American Society of Anesthesiologists (ASA) physical status II-III
* Male patients aged 65 years or younger
* Undergoing lobectomy for the first time
* High nicotine dependence, confirmed by the Fagerström Test for Nicotine Dependence (FTND) with an FTND score of 6 or higher
* No history of substance abuse and no recent use of analgesic medications (e.g., opioids or non-steroidal anti-inflammatory drugs) prior to surgery
* Able to understand the procedure for patient-controlled intravenous analgesia (PCIA) and able to complete the study assessment scales

Exclusion Criteria

* History of mental illness or cognitive disorder; or currently receiving antidepressant treatment and unable to cooperate with examinations and assessments
* Bradycardia (heart rate 50 beats/min or lower) or second- or third-degree atrioventricular block
* Body mass index (BMI) greater than 30 kg/m²
* Use of analgesics, sedatives, beta-blockers, or alpha-2 agonists prior to surgery
* Required reoperation due to serious postoperative complications (e.g., bleeding)
* Severe cardiovascular, cerebrovascular, hepatic, or renal disease, resulting in inability to remove the endotracheal tube after surgery or inability to use the analgesia pump correctly
* Failure to abstain from smoking for at least 2 weeks prior to surgery

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Movement-evoked pain intensity (VAS 0-10) within 48 hours after surgery | Within 48 hours after surgery (assessed at 4, 8, 12, 24, and 48 hours after surgery; primary endpoint is the mean VAS across all assessments during the first 48 hours after surgery).
  Pain during standardized movement (deep breathing/cough or turning in bed) measured on a 10-cm visual analog scale (0=no pain, 10=worst imaginable pain). Trained nurses record scores at each time point. Higher scores indicate worse pain. The primary analysis compares groups on the mean of all movement VAS values collected from 0-48 h postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenyang Chest Hospital, Department of Anesthesiology, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No